CLINICAL TRIAL: NCT03842332
Title: Resilience in Action: Building Resilience and Appropriate Independence in Young Adults With Autism
Brief Title: Building Resilience and Appropriate Independence in Young Adults With Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Golden Gate Regional Center (Unknown); The Arc San Francisco (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P0527544; R21MH115375 (NIH)
Record Dates: First submitted 2018-10-04; First posted 2019-02-15 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This project utilizes an intention to treat, wait-list cross over design of individuals who agree to participate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilience Training (Experimental): This group will participate in the 12 week Life Skills and Resilience Program that includes vocational skills and adult skills important for an adult in society. Participants will also receive standard case management plus resiliency-focused support to encourage family and young adult interaction with professionals and peers. Case managers will then utilize a resiliency framework for their interaction with the participant.
  Interventions: Behavioral: Life Skills and Resilience Program
- Standard Care (No Intervention): This group will receive case management referral to community training programs when requested by family, or need (as identified by case worker). Standard case management includes intake includes housing counseling, case management with mental health and behavioral services, and referral to day programs as needed and identified by case management

INTERVENTIONS:
Behavioral: Life Skills and Resilience Program — The 12 week life skills course includes resiliency modules that complement the strengths of participants as they progress toward the development and achievement of personal goals. The first module of the intervention engages youth through a caring/supportive relationship that sets these expectations. Activities are designed to support youth in identifying their existing strengths/skills. The second module explores, with youth, how they can apply and build upon their strengths/skills in the pursuit of self-generated goals. The third module is dedicated to building upon key problem solving skills that are especially important for young adults with autism, including conflict resolution and the management of stressors. The fourth module builds leadership capacity and self-advocacy skills.
  Arms: Resilience Training

SUMMARY:
This study evaluates the effects of a 12-week life-skills resilience curriculum for young adults with autism. The project utilizes a wait-list crossover design and compares the intervention to standard care.

DETAILED DESCRIPTION:
As young adults with autism spectrum disorder (YAASD) transition out of the academic supports provided by school, these young adults experience a degradation of social skills over time. This has led to poor academic, educational and health outcomes. YAASD require continuous and ongoing skill development in order to maximize their potential; however, there are few services available to adults with autism to develop and maintain their skills. While interventions exist in early childhood, mid-childhood and adolescence, few programs have been focused on the young adult with autism. Resilience in Action (RiA), is a research study, performed and delivered in the community setting, which seeks to develop supports to address the 'adult world' needs of young adults with autism exiting out of secondary education.

The investigators propose to develop this program through three specific aims. In the first aim, the investigators propose in-depth interviews with adults with autism and/or their families and service providers to better understand barriers and facilitators to "adult living" after graduating out of the school system. In the second aim, the investigators will use the information gained from Aim 1 to develop a 12-week curriculum integrating a resilience framework and methodologies into a community adult life skills program for persons with disabilities. A trained transition curriculum expert who had developed transition curriculum for youth with autism spectrum disorder in our local school district will assist in this "adult" curriculum to fill gaps that exist in the school district curriculum. As part of the infrastructure and support for this pilot, the investigators will generate a protocol for the participant's existing case manager to help support youth and families after the curriculum is completed. The third aim is to then pilot test RiA on 30 young adults with autism who have recently graduated from the secondary education system. Through an iterative program evaluation, the investigators will further hone the intervention and adapt the program to different levels of disability and learning styles. The investigators will measure characteristics of those who were successfully engaged in the program and measure outcomes such as socialization, quality of life, vocational/social activities and self-efficacy. Through this research the investigators will have developed a final protocol for a resiliency course to be tested in a larger clinical trial to see how this type of curriculum can improve longer term social and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to high functioning autism spectrum disorder, defined as an SRS T-score less than 75
* Participants must be able to participate in a one hour class with nine other participants and be able to interact with participants and the teacher without support.
* Completing the high school transition program or have exited the school system within the last three years

Exclusion Criteria:

* Non-English speaking
* Unable to consent
* Wards of the state
* Incarcerated.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Baseline Resilience at 3-6 months | Baseline & 3-6 months
  Resilience Scale (RS) developed by Wagnild and Young (1990)
  * Personal competence and acceptance of self and life, which measures the construct of resilience.
  * Adapted for 2nd and 5th grade reading level
  * Possible scores range from 25 to 175 with higher scores reflecting higher resilience
Change in Baseline General Family Functioning at 3-6 months | Baseline & 3-6 months
  McMaster Family Assessment Device (FAD), General Functioning Subscale
  * The General Functioning Subscale ranges from 1 to 4 with higher scores indicating worse levels of family functioning.
  * A score of 2.00 or above indicates problematic family functioning.
Change in Baseline Self Efficacy at 3-6 months | Baseline & 3-6 months
  PROMIS® A person's belief in his/her capacity to manage functioning and have control over meaningful events.
Change in Baseline Pediatric Quality of Life at 3-6 months | Baseline & 3-6 months
  Pediatric Quality of Life Inventory (PedsQL) 4.0 Generic Core Scales
  * Validated quality of life measure that has been developed across different developmental ages and adults
  * Scale ranges from 0 to 100 and higher scores indicate better Health-Related Quality of Life
  * Four sub-scales include Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning
  * Total Scale Score is the mean computed as the sum of all the items over the number of items answered on all the Scales
Change in Baseline Satisfaction with Social Roles at 3-6 months and Activities (v2.0) | Baseline & 3-6 months
  PROMIS Satisfaction with Social Roles and Activities
  * Measures satisfaction with performing one's usual social roles and activities (e.g., "I am satisfied with my ability to participate in family activities")
  * Raw scores (ranging from 6 to 40) are converted to T-scores with a mean of 50 and standard deviation of 10
  * A higher PROMIS T-score represents greater satisfaction with social roles and activities.

SECONDARY OUTCOMES:
Change in Baseline Employment Status | Baseline & 3-6 months
  Percentage of study participants employed

CONTACTS AND LOCATIONS:
Overall Officials: Megumi Okumura, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- The Arc, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No